CLINICAL TRIAL: NCT04133961
Title: Intraoperative Phenylephrine Infusion to Reduce Postoperative Shivering in Lower Segment Caesarean Section
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universiti Kebangsaan Malaysia Medical Centre (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: FF-2019-273
Record Dates: First submitted 2019-10-11; First posted 2019-10-21 (Actual); Last update posted 2020-07-08 (Actual); Status verified 2019-10

CONDITIONS: Postoperative Shivering
Keywords: Phenylephrine; Spinal anaesthesia
MeSH Terms: interventions — Phenylephrine; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Phenylephrine) (Experimental): Phenylephrine infusion started immediately after administration of spinal block
  Interventions: Drug: Phenylephrine
- Group B (Saline) (Placebo Comparator): Normal saline infusion started immediately after administration of spinal block
  Interventions: Drug: Normal saline

INTERVENTIONS:
Drug: Phenylephrine — Phenylephrine infusion 0.3ml/kg/hour (equivalent to 0.5mcg/kg/min, phenylephrine dilution is 100mcg/ml in 20ml syringe)
  Arms: Group A (Phenylephrine)
Drug: Normal saline — Normal saline infusion 0.3ml/kg/hour (normal saline in 20ml syringe)
  Arms: Group B (Saline)

SUMMARY:
Assessment of whether and how phenylephrine infusion reduces postoperative shivering in spinal anaesthesia.

DETAILED DESCRIPTION:
This study aims to evaluate whether phenylephrine infusion can reduce postoperative shivering among patients scheduled for elective lower segment caesarean section under spinal anaesthesia.

ELIGIBILITY:
Inclusion Criteria:

* More than 18 years of age
* American Society of Anesthesiologists (ASA) II patients
* Patients with singleton pregnancy who are scheduled to undergo elective lower segment caesarean section under spinal anaesthesia

Exclusion Criteria:

* Patients with contraindication to phenylephrine
* Patients with evidence of fever or infection, or hypothermia preoperatively
* BMI ≥ 40
* Height <150cm

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Patients who are planned for elective lower segment caesarean section
Enrollment: 118 (Actual)
Dates: Start 2019-06-12 (Actual); Primary Completion 2019-12-01 (Actual); Study Completion 2020-01-01 (Actual)

PRIMARY OUTCOMES:
Presence and intensity of shivering | 2 hours
  Any presence of shivering intraoperatively is recorded. The intensity of shivering is recorded based on the Bedside Shivering Assessment Scale (BSAS) with a scoring of 0-3 (0 = no shivering, 1 = shivering localised to neck and/or thorax, 2 = shivering involves gross movement of upper extremities, 3 = shivering involves gross movements of the trunk, upper and lower extremities).

SECONDARY OUTCOMES:
Change in patient's core and skin temperature | 2 hours
  Patient's core (tympanic membrane) and skin (forehead) temperature is measured using an infrared thermometer.

CONTACTS AND LOCATIONS:
Overall Officials: Syarifah Noor Nazihah Sayed Masri, MD, Principal Investigator — Anaesthesiologist
Locations (1):
- Pusat Perubatan Universiti Kebangsaan Malaysia, Kuala Lumpur, Malaysia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ikeda T, Ozaki M, Sessler DI, Kazama T, Ikeda K, Sato S. Intraoperative phenylephrine infusion decreases the magnitude of redistribution hypothermia. Anesth Analg. 1999 Aug;89(2):462-5. doi: 10.1097/00000539-199908000-00040. PMID 10439767
- [Background] Ro Y, Huh J, Min S, Han S, Hwang J, Yang S, Kim DK, Kim C. Phenylephrine attenuates intra-operative hypothermia during spinal anaesthesia. J Int Med Res. 2009 Nov-Dec;37(6):1701-8. doi: 10.1177/147323000903700605. PMID 20146867
- [Background] Hilton EJ, Wilson SH, Wolf BJ, Hand W, Roberts L, Hebbar L. Effect of Intraoperative Phenylephrine Infusion on Redistribution Hypothermia During Cesarean Delivery Under Spinal Anesthesia. J Clin Anesth Manag. 2016 Jan;1(1):10.16966/2470-9956.103. doi: 10.16966/2470-9956.103. Epub 2015 Dec 19. PMID 32500108
- [Background] Badjatia N, Strongilis E, Gordon E, Prescutti M, Fernandez L, Fernandez A, Buitrago M, Schmidt JM, Ostapkovich ND, Mayer SA. Metabolic impact of shivering during therapeutic temperature modulation: the Bedside Shivering Assessment Scale. Stroke. 2008 Dec;39(12):3242-7. doi: 10.1161/STROKEAHA.108.523654. Epub 2008 Oct 16. PMID 18927450